CLINICAL TRIAL: NCT05072678
Title: Clinical and Radiological Evaluation of Two Mastoid Filling Products in Patients With Cholesteratoma.
Brief Title: Clinical and Radiological Evaluation of Two Mastoid Filling Products
Acronym: MASTOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0018 (MASTOS)
Record Dates: First submitted 2021-04-29; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-04

CONDITIONS: Prospective Study
Keywords: osteoingration; surgery; cholesteatome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to compare, the osseous density in the mastoid of two products used to obliterate the mastoid during surgery for cholesteatoma

DETAILED DESCRIPTION:
Primary objective: To compare the radiological aspect in the petrous bone of two obliteration products in adults, one year after surgery (Bioactive Glass S53P4 and biological Hydroxy apatite) secondary objective : To evaluate the cutaneous and the inner ear tolerance of bioactive glass S53P4 and biological hydroxy apatite when used in the mastoid and epitympanic obliteration for chronic otitis surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult with cholesteatoma surgery Accepting the protocol and the radiological follow-up

Exclusion Criteria:

* patient less than 18 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cholesteatoma surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-04-25 (Actual); Primary Completion 2022-04-25 (Estimated); Study Completion 2023-04-25 (Estimated)

PRIMARY OUTCOMES:
Hounsfield Unit | one year
  The attenuation and osseointegration of the BG granules:
  The quantitative analysis included bone attenuation measurements (in Hounsfield units, HU) in the circular region of interest (34mm2) of BGand of surrounding cortical bone and otic capsule using the otic capsule adjacent to the LSCC and the posterior fossa dural plate (DP)

SECONDARY OUTCOMES:
decibel | one year
  Auditory level pre and postoperative evaluation clinical
decibel | one year
  audiological evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU De Brest, Brest, France